CLINICAL TRIAL: NCT05810155
Title: Delayed Elective Surgery in Inflammatory Bowel Disease - a Health Economic Analysis Including Quality of Life
Brief Title: Delayed Surgery in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bjarne Melvas, MD, Sahlgrenska University Hospital
Other Study IDs: 2022-05975-01
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Quality of Life; Surgery
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time waiting for surgery: This group includes all patients with IBD who are waiting for elective surgery and was put on the waiting list 2017-2021 at Sahlgrenska University Hospital.
- Operated: This group includes patients with IBD who was operated with elective surgery 2017-2021 at Sahlgrenska University Hospital.

SUMMARY:
The timing of elective surgery in inflammatory bowel disease (IBD) may be crucial according to progression of the disease. In most cases, medical treatment has failed when surgery is discussed. If treatment with surgery then is delayed, complications may arise, such as fistula, severe inflammation with risk of perforation or stenosis, nutrition problems i.e. This may affect quality of life, and also make the surgery more complicated, with higher risk of per- and postoperative complications.

The COVID-19 pandemic led to a shift in resources where elective surgery has been postponed. The waiting time for elective surgery for IBD-patients at Sahlgrenska University Hospital/Östra is still affected which might have impact on patient health outcomes as well as health economics, due to the risk of complications and need of emergency and planned care while waiting for surgery.

The primary object is to evaluate how long an IBD patient can wait for surgery before affecting health economy and quality of life. In the operation program Orbit, we identify all patients with ulcerative colitits (UC) and Crohn´s disease (CD) that stands in line for elective surgery (not including dysplasia/cancer). The date when operation was decided is registered including time of delay. Patient characteristics are registered in CRF, including diagnosis, age and reason for scheduled surgery. Number of hospital visits (planned/emergency visits) are registered during time of waiting for surgery. Days of sick leave is registered from the Swedish Social Insurance Agency. Questionnaires are sent to the patients for quality of life and bowel function (EQ5D and Short Health Scale).

The primary endpoint in the first manuscript is how health economics is affected by the delay of elective care in IBD-patients, due to complications and extensive need of hospital visits while waiting for surgery, costs of medical material (stoma bandage i.e), costs of medical treatment and sick leave rates, including quality of life. Patients who have been operated for IBD will form the control group and comparison will be made in terms of complications, hospital visits, costs of medical material and medical treatment and sick leave rates, as well as quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel Disease
* Minimum 18 years old
* Planned surgery/operated since 2017-2021 at Sahlgrenska University Hospital

Exclusion Criteria:

* cancer surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with IBD with planned elective surgery or operated 2017-2021
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
How is health economy including quality of life affected when surgery is delayed? | 2023/2024
  Regarding patients with IBD.

SECONDARY OUTCOMES:
Socioeconomic differences in delayed surgery | 202472025
Does waiting for surgery affect the result? | 2026
  Complications, failures.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hermanson, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Sweden